CLINICAL TRIAL: NCT01333787
Title: A Controlled, Randomized, Double-blind Trial to Evaluate the Effect of a Dietary Fiber Mixture During Maintenance Treatment and on Colonic Transit Time in Constipated Pediatric Patients
Brief Title: Dietary Fiber Mixture in Constipated Pediatric Patients
Acronym: MIXFIBER
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Collaborators: Mauro Batista de Morais (Unknown); Soraia Tahan (Unknown); Mauro Sérgio Toporovski (Unknown); Clarice Blaj Neufeld (Unknown); Thabata Koester Weber (Unknown)
Responsible Party: Mauro Batista de Morais, Federal University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FiberCCF - EPM2
Record Dates: First submitted 2011-04-11; First posted 2011-04-12 (Estimated); Last update posted 2011-04-12 (Estimated); Status verified 2010-12

CONDITIONS: Constipation
Keywords: dietary fiber; clinical trial; constipation; children
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dietary Fiber Mixture (Active Comparator): The dietary fiber mixture was composed of six different types of fibers. It was used for treatment of chronic constipation in children.
  Interventions: Dietary Supplement: Dietary Fiber Mixture
- Maltodextrine (Placebo Comparator): Blinded control group
  Interventions: Dietary Supplement: Dietary Fiber Mixture

INTERVENTIONS:
Dietary Supplement: Dietary Fiber Mixture — During the four weeks the patients received fiber mixtures (intervention) or maltodextrine as the placebo. The fiber mixture was composed of six different types of fibers: 10.5% fructooligosaccharides, 12.5% inulin, 24% Arabic gum, 9% resistant starch, 33% Soya polysaccharide e 12% cellulose.
  The dose was defined in accordance with the child's body weight: 6.3 grams of fiber supplement, which corresponds to 4.8 g of fiber, or placebo(1 table spoon) twice per day, diluted in 200 mL of a milky chocolate drink for children weighing up to 18 kg; 12.6 grams of fiber supplement, which corresponds to 9.6 g of fiber, or placebo (2 table spoons) twice per day, diluted in 200 mL of a milky chocolate drink for children weighing more than 18 Kg.
  Other Names: Stimulance

SUMMARY:
The purpose this study was to to evaluate the therapeutic effect of a fibers mixture in the treatment of chronic constipation and on the colonic transit time in children.

DETAILED DESCRIPTION:
In spite of an increase in the consumption of fibers being indicated for the treatment of constipation, few clinical trails have evaluated its efficiency. In the majority of prior studies only the effect of a single type of fiber was evaluated. Each type of fiber presents a particular characteristic, which determines its action mechanism and performance in different parts of the colon. Therefore, theoretically, greater effectiveness could well be observed when different types of fibers are associated into a single product for fiber supplementation.

A randomized, parallel, double-blind, controlled was performed to evaluate the effect of a dietary fiber mixture in constipated pediatric patients.

Children aged between 4 and 12 years were included in the study and the initial diagnosis of functional chronic constipation was made in accordance with the Rome III criteria. The children having attended the Pediatric Gastroenterology Ambulatory of the Federal University of Sao Paulo and the Santa Casa de Misericórdia hospital in Sao Paulo city. All of the children were undergoing constipation maintenance treatment with the use of a laxative in a dosage less than 1.0 ml/Kg for milk of magnesia, mineral oil or lactulose or less than 0.5 g/Kg for polyethylene glycol 3350.

ELIGIBILITY:
Inclusion Criteria:

* Children aged between 4 and 12 years;
* Maintenance treatment using low dose of laxative;
* A family with the socio-economic culture that would make it possible to carry out the procedures of the study's protocol.

Exclusion Criteria:

* Children with organic cause constipation such as Hirschsprung disease, cerebral paralysis, anorectal and spinal medulla abnormalities and metabolic illnesses;
* The regular use of a fiber supplement during the 4 weeks prior to admission;
* The use of medications that would cause constipation;
* Absence of a fixed or mobile telephone in order to make contact.

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 54 (Actual)
Dates: Start 2008-02; Primary Completion 2009-01 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Clinical response - Therapeutic success | 4 weeks
  The primary outcome result measurement was the therapeutic success. This therapeutic success was considered when the patient demonstrated daily evacuations or had interposing days of pasty consistency, without pain or difficulty and the absence of fecal incontinence during the 4 weeks of intervention, without the need of using a laxative or rectal enema.

SECONDARY OUTCOMES:
Frequent daily evacuations, format and consistency of the feces, total and segmental transit time | 4 weeks
  The format and consistency of the feces was evaluated in accordance with the Bristol Stool Form Scale (stool are rated based on water content of the feces, with 1 meaning hard stools to 7 meaning liquid stools).
  The colonic transit time was evaluated during the study's final week by way of the method proposed by Bouchoucha et al. (1992).

CONTACTS AND LOCATIONS:
Locations (1):
- UNIFESP - Pediatric Gastroenterology Ambulatory, São Paulo, São Paulo, Brazil